CLINICAL TRIAL: NCT04563598
Title: The Effects of an Intensive Lifestyle Intervention for Type 2 Diabetes on Employment, Earnings, and Retirement
Brief Title: The Effects of an Intensive Lifestyle Intervention on Employment, Earnings, and Retirement
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Southern California (Other); Wake Forest University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: UP-16-00706-3; 5R01DK107552 (NIH)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ILI/ Treatment group: This group includes Look AHEAD participants who were initially assigned to the intensive lifestyle intervention (ILI), consented to administrative data linkages, and were successfully linked to Social Security Administration databases.
  Interventions: Behavioral: Intensive lifestyle intervention (ILI)
- DSE/Control group: This group includes Look AHEAD participants who were initially assigned to the diabetes support and education (DSE) control arm, consented to administrative data linkages, and were successfully linked to Social Security Administration databases.
  Interventions: Behavioral: Diabetes support and education (DSE)

INTERVENTIONS:
Behavioral: Intensive lifestyle intervention (ILI) — Lifestyle intervention focused on weight loss through diet and physical activity
  Groups: ILI/ Treatment group
Behavioral: Diabetes support and education (DSE) — Behavioral intervention focused on diabetes support and education
  Groups: DSE/Control group

SUMMARY:
Starting in 2001, the Look AHEAD study randomized patients with type 2 diabetes to an intensive lifestyle intervention (ILI) focused on weight loss versus a control group receiving diabetes education ("Diabetes Support and Education," or DSE). The ILI successfully reduced weight, improved diabetes control, and functional status, among other outcomes. In this study, the investigators will compare employment, earnings, and retirement between the ILI and the control group during and after the intervention period (2001-2018).

DETAILED DESCRIPTION:
Starting in 2001, the Look AHEAD study randomized 5145 patients with type 2 diabetes to an intensive lifestyle intervention (ILI) focused on weight loss versus a control group receiving diabetes education ("Diabetes Support and Education," or DSE).The Look AHEAD study tested whether participants with type 2 diabetes assigned to an intensive lifestyle intervention (ILI) for weight loss exhibited reductions in cardiovascular morbidity and mortality, relative to a control group receiving usual care and diabetes support and education. During the 12-year intervention period, the ILI led to persistent reductions in weight, waist circumference, and hemoglobin A1c and improvements in physical fitness, among other clinical benefits. After the conclusion of the intervention in 2012, participants were consented to be linked with administrative data. The investigators attempted to link 3188 consenting participants with Social Security Administration databases. Of these, the investigators were able to successfully link 3093 participants. In this study, the investigators will compare employment, earnings, and retirement between the ILI and the control group during and after the intervention period (2001-2018). The investigators will determine ILI-versus-control differences in employment, earnings, and retirement in each year after randomization, relative to a pre-randomization assessment period. The investigators will also investigate ILI-versus-control differences in cumulative years of employment and earnings after randomization which occurred between 2001-2004. The investigators will use multivariate regressions controlling for baseline participant characteristics and clinic site and also survival analyses that estimate whether the time until retirement differs between the ILI and control groups.

ELIGIBILITY:
(Note: age limits above are at time of randomization, which occurred between 2001-2004)

Inclusion Criteria:

* Look AHEAD participation: met age requirements and other criteria at time of study enrollment which occurred between 2001-2004 (as noted in Look AHEAD Research Group (2013))
* Consented to administrative data linkages
* Provided individual identifiers that could be linked with Social Security Administration databases
* Were successfully linked to Social Security Administration data

Exclusion Criteria:

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes Look AHEAD participants who consented to administrative data linkages, provided individual identifiers that could be linked with Social Security Administration data, and were successfully linked to Social Security Administration data.
Sampling Method: Non-Probability Sample
Enrollment: 3091 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Employed (any earnings from employment or self-employment) by study year (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on earnings
Total earnings from employment and/or self-employment by study year (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on earnings; earnings for unemployed study participants will be captured as zeros.

SECONDARY OUTCOMES:
Retired (any Social Security retirement entitlement/election) by study year (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on retirement entitlement/election
Total earnings from employment and/or self-employment by study year (excluding unemployed study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on earnings
Total person-years from randomization to retirement (all study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on retirement entitlement/election
Total person-years employed since randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on earnings
Ever employed (any earnings from employment or self-employment) after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on earnings
Total earnings from employment and/or self-employment since randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on earnings
Ever received Supplemental Security Income (SSI) benefits at age 65 since randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data indicating SSI benefits and SSI eligibility.

OTHER OUTCOMES:
Number of employers (unique employer IDs) per study year (excluding unemployed study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on employers
Started a new job (new employer ID) by study year (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on employment
Started a new job (new employer ID) by study year (excluding unemployed study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on employment
Received any Supplemental Security Income (SSI) benefits at age 65 since randomization (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data indicating SSI benefits and SSI eligibility
Received any self-employment income by study year (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on earnings
Received any income from pensions or distributions from retirement accounts by study year (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on earnings
Total compensation (from employment, self-employment, pensions, and distributions from retirement accounts (all study participants) | 12-month intervals relative to randomization occurring between 2001-2018
  This measure is based on Social Security Administration data on compensation
Ever retired after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on retirement entitlement/election
Ever worked past minimum retirement age (partial benefits, age 62; excluding unemployed study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on earnings
Ever worked past minimum retirement age (full benefits, age 65 or 66 depending on date of birth; excluding unemployed study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on earnings
Total compensation (from employment, self-employment, pensions, and distributions from retirement accounts) after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2018
  This measure is based on Social Security Administration data on compensation
Ever employed (any earnings from employment and/or self-employment) during first 10 years after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2014
  This measure is based on Social Security Administration data on earnings
Total person-years employed (any earnings from employment and/or self-employment) during first 10 years after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2014
  This measure is based on Social Security Administration data on earnings
Total earnings (from employment and/or self-employment) during first 10 years after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2014
  This measure is based on Social Security Administration data on earnings
Total compensation (from employment, self-employment, pensions, and distributions from retirement accounts) during first 10 years after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2014
  This measure is based on Social Security Administration data on compensation
Ever retired during first 10 years after randomization (all study participants) | From initial randomization (occurred between 2001-2004) through 2014
  This measure is based on Social Security Administration data on retirement entitlement/election

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Huckfeldt, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No
Use of Social Security Administration data is restricted under a data use agreement between the Social Security Administration and Wake Forest University.

REFERENCES:
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131